CLINICAL TRIAL: NCT03162081
Title: Medication Misuse and Dependence in Elderly Patients
Brief Title: Medication Misuse and Dependence Among Elderly
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: King's College London (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Christofer Lundqvist, Principal investigator, University Hospital, Akershus
Other Study IDs: NRC256431WP2
Record Dates: First submitted 2017-05-03; First posted 2017-05-22 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Mild Cognitive Impairment; Elderly; Substance-Related Disorders
Keywords: addiction; cognition; impulsivity; neuropsychology; prescription drug misuse; dependence
MeSH Terms: conditions — Cognitive Dysfunction; Substance-Related Disorders; Behavior, Addictive; Impulsive Behavior; Prescription Drug Misuse | interventions — Medication Errors; Comorbidity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Users: Elderly patients who use prescription benzodiazepines/Z-hypnotics or opiates
  Clinical interview, Substance misuse screening, EuroQol five dimensional health-related quality of life questionnaires (EQ-5D), Impulsivity screening, Cognitive screening, Functional tests, Cognistat Neurobehavioural cognitive status examination (Cognistat), Neuropsychological profiling, Medication use, Comorbidity
  Interventions: Diagnostic Test: Substance misuse screening; Diagnostic Test: EQ-5D; Diagnostic Test: Impulsivity screening; Diagnostic Test: Cognitive screening; Diagnostic Test: Functional tests; Diagnostic Test: Cognistat; Diagnostic Test: Neuropsychological profiling; Other: Clinical interview; Other: Medication use; Other: Comorbidity
- Non-users: Age and gender matched controls not using the above
  Clinical interview, Substance misuse screening, EuroQol five dimensional health-related quality of life questionnaires (EQ-5D), Impulsivity screening, Cognitive screening, Functional tests, Cognistat Neurobehavioural cognitive status examination (Cognistat), Neuropsychological profiling, Medication use, Comorbidity
  Interventions: Diagnostic Test: Substance misuse screening; Diagnostic Test: EQ-5D; Diagnostic Test: Impulsivity screening; Diagnostic Test: Cognitive screening; Diagnostic Test: Functional tests; Diagnostic Test: Cognistat; Diagnostic Test: Neuropsychological profiling; Other: Clinical interview; Other: Medication use; Other: Comorbidity
- Screening group: Patients over 65 admitted to hospital as in-patients
  Clinical interview, Substance misuse screening, EuroQol five dimensional health-related quality of life questionnaires (EQ-5D), Impulsivity screening, Cognitive screening, Functional tests, Medication use, Comorbidity
  Interventions: Diagnostic Test: Substance misuse screening; Diagnostic Test: EQ-5D; Diagnostic Test: Impulsivity screening; Diagnostic Test: Cognitive screening; Diagnostic Test: Functional tests; Other: Clinical interview; Other: Medication use; Other: Comorbidity

INTERVENTIONS:
Diagnostic Test: Substance misuse screening — Diagnostic and Statistical manual of mental disorders, version 4 (DSM-IV)/MINI-international Neuropsychiatric interview (MINI interview) for Diagnostics of dependence, additional questions for DSM-V classification, severity of dependence scale (SDS)
Diagnostic Test: EQ-5D — Health related Quality of life
Diagnostic Test: Impulsivity screening — Barratts impulsivity test v. 11, Behavioural inhibition/behavioural activation test
Diagnostic Test: Cognitive screening — Minimental state examination (MMSE), Hospital anxiety and depression scale (HADS), Trail-making test, clock drawing test
Diagnostic Test: Functional tests — Timed up and go (TUG), Single leg balancing test (SLB)
Diagnostic Test: Cognistat — Assessment of cognitive domains
  Groups: Non-users; Users
Diagnostic Test: Neuropsychological profiling — Controlled Oral Word Association Test, Categorical fluency tests, Wechsler Adult Intelligence Scale, Color-Word Interference Test (CWIT) from the Delis-Kaplan Executive Function test
  Groups: Non-users; Users
Other: Clinical interview — Interview for sociodemographics, utilisation of health care, economic varables, The De Jong Gierveld Loneliness Scale
Other: Medication use — Detailed screen of used medications, interactions, side effects in electronic patient registry
Other: Comorbidity — Charlson comorbidity index and Cumulated illness rating scale (CIRS) based on electronic patient registry

SUMMARY:
The project focuses on investigating problematic medication use, especially overuse of potentially addictive drugs among the elderly.

The investigators aim firstly to develop and validate instruments for detecting and describing behavioral aspects and consequences of dependence on, and misuse of, prescription medication among elderly.

In addition to evaluating diagnostic utility of screening instruments, the investigators aim to identify and report characteristics, risk factors and consequences of medication misuse and dependence among the elderly.

DETAILED DESCRIPTION:
Elderly represent a particularly vulnerable group with many contributing factors including age-related multifactorial morbidity, cognitive function, polypharmacy, dependence and multiple prescribers with suboptimal communication. Centrally active pain killers and sedative/hypnotic medications give increased risk of addiction, adverse drug events, reduced physical and/or cognitive function.

The project comprises diagnostic accuracy, descriptive screening, cross-sectional and case-control studies, with aims to: i) assess diagnostic utility of instruments for elderly patients; ii) describe risk factors for medication misuse and dependence; iii) describe consequences of the use of centrally active medications among elderly compared to a control population.

Moreover, the investigators aim to examine the association between medication misuse and changes in cognitive function, focusing on deficits in specific domains of cognition. An additional aim is to explore the possibility of dissociating such cognitive changes from other causes of mild cognitive impairment (MCI) associated with development of dementia.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to geriatric or Neurology dept of hospital during inclusion time

Exclusion Criteria:

* MMSE < 21,
* diagnosis of pre-existing severe depression or psychotic disease,
* pre-existing dementia diagnosis,
* new pain requiring start-up of central pain killers not previously used,
* Palliative treatment.
* Insufficient Norwegian language
* Serious visual disturbance and hearing impairment
* Strongly reduced general health precluding partcipation in interview and questionnaires

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All admitted elderly 65-90 years of age are screened, for case-control age and gender-matched pairs of Users and non-users will in addition be examined in depth with neuropsychological tests
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Dependence y/n | Within 2 weeks of admission
  DSM-IV defined substance dependence assessed by MINI interview
Medication misuse y/n | Past year prior to in-hospital stay (data collected within 2 weeks of admission)
  Use of any of: opiates/benzodiazepine/Z-hypnotics >5 days per week for >3 months

SECONDARY OUTCOMES:
MCI - Mild cognitive impairment | Within 2 weeks of admission
  Defined by MMSE < 26
MMSE | Within 2 weeks of admission
  Numerical score of cognitive function
COGNISTAT | Within 2 weeks of admission
  Cognitive profile
EQ-5D | Within 2 weeks of admission
  Quality of life
BIS-11 | Within 2 weeks of admission
  Impulsivity score
BIS/BAS score | Within 2 weeks of admission
  Behavioura inhibition/activation score
TUG | Within 2 weeks of admission
  Functional test score (time in secs)
SLB | Within 2 weeks of admission
  Functional test score (time in secs)
Neuropsychological profiles | Within 2 weeks of admission
  Tests as listed
Use of addictive medication y/n | Within 2 weeks of admission
  Prescription use of any of the following: opiates, benzodiazepines, Z-hypnotics
No of days of use of defined addictive medications/month | Within 2 weeks of admission
  No. days of use of any of the following: opiates, benzodiazepines, Z-hypnotics
No. of possible side effects | Within 2 weeks of admission
  No. possible side effects of any of the following: opiates, benzodiazepines, Z-hypnotics
No. of possible serious interactions | Within 2 weeks of admission
  No. possible serious interactions of any of the following: opiates, benzodiazepines, Z-hypnotics
No.of inappropriate medications for elderly at admission | Within 2 weeks of admission
  No.of inappropriate medications as defined by NORGEP criteria (Norwegian general practice criteria)
No.of inappropriate medications for elderly during in-hospital stay | Within 2 weeks of admission
  No.of inappropriate medications as defined by NORGEP criteria
No.of inappropriate medications for elderly at discharge | Within 2 weeks of admission
  No.of inappropriate medications as defined by NORGEP criteria
No.of inappropriate medications for elderly at admission | Within 2 weeks of admission
  No.of inappropriate medications as defined by STOPP criteria (Screening tool of older patients prescriptions)
No.of inappropriate medications for elderly during in-hospital stay | Within 2 weeks of admission
  No.of inappropriate medications as defined by STOPP criteria
No.of inappropriate medications for elderly at discharge | Within 2 weeks (index stay may in some cases be somewhat longer)
  No.of inappropriate medications as defined by STOPP criteria
Substance use disorder | Within 2 weeks
  DSM-IV criteria assessed through additional questions to MINI interview

OTHER OUTCOMES:
Mortality | 2 years
  Crude mortality from patient registry data
Mortality | 5 years
  Crude mortality from patient registry data
Readmission rate | 5 years
  Number of readmissions after index admission
Total readmission days | 5 years
  Total number of readmission days

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn Rugkåsa, PhD, Study Director — Coordinator of overall research program
Locations (1):
- Akershus University Hospital, Lørenskog, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bjelkaroy MT, Simonsen TB, Siddiqui TG, Cheng S, Grambaite R, Benth JS, Lundqvist C. Mortality and health-related quality of life in older adults with long-term use of opioids, z-hypnotics or benzodiazepines: a prospective observational study at 5 years follow-up. BMJ Open. 2024 Feb 21;14(2):e079347. doi: 10.1136/bmjopen-2023-079347. PMID 38387984
- [Derived] Bjelkaroy MT, Simonsen TB, Siddiqui TG, Halset S, Cheng S, Grambaite R, Benth JS, Gerwing J, Kristoffersen ES, Lundqvist C. Brief Intervention as a Method to Reduce Z-Hypnotic Use by Older Adults: Feasibility Case Series. JMIR Form Res. 2024 Feb 8;8:e51862. doi: 10.2196/51862. PMID 38329779
- [Derived] Bjelkaroy MT, Benth JS, Simonsen TB, Siddiqui TG, Cheng S, Kristoffersen ES, Lundqvist C. Measuring pain intensity in older adults. Can the visual analogue scale and the numeric rating scale be used interchangeably? Prog Neuropsychopharmacol Biol Psychiatry. 2024 Mar 2;130:110925. doi: 10.1016/j.pnpbp.2023.110925. Epub 2023 Dec 22. PMID 38143014
- [Derived] Siddiqui TG, Bjelkaroy MT, Cheng S, Kristoffersen ES, Grambaite R, Lundqvist C. The effect of cognitive function and central nervous system depressant use on mortality-A prospective observational study of previously hospitalised older patients. PLoS One. 2022 Mar 3;17(3):e0263024. doi: 10.1371/journal.pone.0263024. eCollection 2022. PMID 35239678
- [Derived] Bjelkaroy MT, Cheng S, Siddiqui TG, Benth JS, Grambaite R, Kristoffersen ES, Lundqvist C. The association between pain and central nervous system depressing medication among hospitalised Norwegian older adults. Scand J Pain. 2021 Dec 16;22(3):483-493. doi: 10.1515/sjpain-2021-0120. Print 2022 Jul 26. PMID 34913326
- [Derived] Siddiqui TG, Cheng S, Gossop M, Kristoffersen ES, Grambaite R, Lundqvist C. Association between prescribed central nervous system depressant drugs, comorbidity and cognition among hospitalised older patients: a cross-sectional study. BMJ Open. 2020 Jul 27;10(7):e038432. doi: 10.1136/bmjopen-2020-038432. PMID 32718926
- [Derived] Cheng S, Siddiqui TG, Gossop M, Kristoffersen ES, Lundqvist C. Sociodemographic, clinical and pharmacological profiles of medication misuse and dependence in hospitalised older patients in Norway: a prospective cross-sectional study. BMJ Open. 2019 Sep 5;9(9):e031483. doi: 10.1136/bmjopen-2019-031483. PMID 31492795
- [Derived] Cheng S, Siddiqui TG, Gossop M, Kristoffersen ES, Lundqvist C. The Severity of Dependence Scale detects medication misuse and dependence among hospitalized older patients. BMC Geriatr. 2019 Jun 24;19(1):174. doi: 10.1186/s12877-019-1182-3. PMID 31234786